CLINICAL TRIAL: NCT01685710
Title: The Use of Glyceryl Trinitrate Patches in Arteriovenous Fistulas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Mr Nick Inston, Consultant Surgeon, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRK4178
Record Dates: First submitted 2012-08-30; First posted 2012-09-14 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Renal Failure
Keywords: Arteriovenous fistula; Patency; GTN patch
MeSH Terms: conditions — Renal Insufficiency; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTN patch (Experimental): GTN patch 5mg, in situ 24hrs
  Interventions: Drug: GTN patch
- Placebo patch (Placebo Comparator): Placebo patch, in situ for 24hrs
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: GTN patch
  Other Names: Minitran 5
  Arms: GTN patch
Drug: placebo comparator — This arm will be a placebo patch to the active drug patch to blind the trial.
  Arms: Placebo patch

SUMMARY:
The aim of the study is to determine whether the application of a glyceryl trinitrate patch (GTN patch) helps arteriovenous fistulas, created for renal dialysis access, mature so that they can be used.

DETAILED DESCRIPTION:
Patients with end stage renal failure on haemodialysis must have a mechanism for achieving access to their vascular system for dialysis. Arteriovenous fistulas (surgically created connections between the artery and vein) are critical for the majority of patients. Not all the fistulas that are created work, a proportion fail early on and need to be revised or an alternative fistula created. A recent multicentre study demonstrated a 40% primary failure rate(1). In an attempt to increase the numbers of fistulae that reach maturation sufficient for dialysis access cannulation some renal centres apply GTN patches to the fistula at the time of surgery. It is thought that this works by increasing the size of the blood vessels and promoting blood flow through them and some preliminary work seems to support this(2).

The evidence for the use of GTN patches in arteriovenous fistula creation is theoretical or based on preliminary work rather than robust evidence. Similarly no evidence exists within the literature to determine the safety and definite efficacy of this procedure in this population. We propose to conduct a double-blinded randomised control trial to answer the study question: does the application of a GTN patch increase the venous outflow diameter post fistula formation and does this result in improved fistula patency.

ELIGIBILITY:
Inclusion Criteria:

* Primary arteriovenous fistulas

  * Brachiocephalic
  * Radiocephalic (both proximal and distal)
* >18 yrs old
* Diabetics and smokers will be eligible for inclusion

Exclusion Criteria:

* All complex vascular access procedures

  * Re-do brachiocephalic and radiocephalic fistulas
  * Brachiobasilic fistulas
  * Prosthetic grafts
* Cardiovascular dysfunction

  * Hypotension (systolic <90)
  * Obstructive Cardiomyopathy
  * Severe Aortic stenosis (gradient >40mmhg)
  * Confirmed myocardial infarction within the last 6 months
* Marked anaemia (Hb<8)
* Migraine
* Medications

  * Sildenafil
  * Pre-existing nitrate use
* Nitrate allergy
* Closed-angle glaucoma
* Chronically raised intra-cranial pressure
* History of hypothyroid disease
* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change to diameter of vein | Initial assessment and 6 weeks after surgery
  At initial assessment of the vein the size will be recorded for later comparison. This will then be re-assessed at 6 weeks post-surgery to allow the change in venous diameter to be assessed.

SECONDARY OUTCOMES:
Number of participants with adverse events | 6 weeks
  Those receiving the active patch will be compared with those receiving the placebo patch for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas G Inston, FRCS, Principal Investigator — University Hospital Birmingham, UK.
Locations (1):
- Queen Elizabeth Hospital, Birmingham., Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Huijbregts HJ, Bots ML, Wittens CH, Schrama YC, Moll FL, Blankestijn PJ; CIMINO study group. Hemodialysis arteriovenous fistula patency revisited: results of a prospective, multicenter initiative. Clin J Am Soc Nephrol. 2008 May;3(3):714-9. doi: 10.2215/CJN.02950707. Epub 2008 Feb 6. PMID 18256379
- [Background] Akin EB, Topcu O, Ozcan H, Ersoz S, Aytac S, Anadol E. Hemodynamic effect of transdermal glyceryl trinitrate on newly constructed arteriovenous fistula. World J Surg. 2002 Oct;26(10):1256-9. doi: 10.1007/s00268-002-6515-1. Epub 2002 Sep 4. PMID 12205547
- [Derived] Field M, McGrogan D, Marie Y, Joinson M, Andujar C, Dutton M, Krishnan H, Hodson J, van Dellen D, Inston NG. Randomized clinical trial of the use of glyceryl trinitrate patches to aid arteriovenous fistula maturation. Br J Surg. 2016 Sep;103(10):1269-75. doi: 10.1002/bjs.10217. Epub 2016 Jul 29. PMID 27470183